CLINICAL TRIAL: NCT02794883
Title: A Phase II, Open Label, Clinical Trial Of Pre-Surgical and Adjuvant Treatment of Recurrent Malignant Glioma With Tremelimumab and Durvalumab (MEDI4736) Alone and in Combination to Determine Immunologic Changes From Treatment
Brief Title: Tremelimumab and Durvalumab in Combination or Alone in Treating Patients With Recurrent Malignant Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: AstraZeneca (Industry); MedImmune LLC (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NU 15C03; STU00202283 (CTRP (Clinical Trial Reporting Program)); NU 15C03 (Other: Northwestern University); P30CA060553 (NIH); NCI-2016-00665 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2016-05-27; First posted 2016-06-09 (Estimated); Results first posted 2022-04-18 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-03

CONDITIONS: Malignant Glioma; Recurrent Glioblastoma
MeSH Terms: conditions — Glioma; Glioblastoma | interventions — durvalumab; Immunoglobulin G; Disulfides; Surgical Procedures, Operative; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment (durvalumab) (Active Comparator): Patients receive durvalumab IV over 1 hour on days 1 and 15. Courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Durvalumab; Other: Laboratory Biomarker Analysis; Procedure: Surgical Procedure
- Treatment (tremelimumab and durvalumab) (Active Comparator): Patients receive tremelimumab IV over 1 hour on day 1 then durvalumab IV over 1 hour on days 1 and 15. Courses repeat every 4 weeks for up to 7 courses. Patients then receive both tremelimumab and durvalumab IV over 1 hour every 12 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Durvalumab; Other: Laboratory Biomarker Analysis; Procedure: Surgical Procedure; Biological: Tremelimumab
- Treatment (tremelimumab) (Experimental): Patients receive tremelimumab IV over 1 hour on day 1. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Procedure: Surgical Procedure; Biological: Tremelimumab

INTERVENTIONS:
Biological: Durvalumab — Given IV
  Other Names: Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736
  Arms: Treatment (durvalumab); Treatment (tremelimumab and durvalumab)
Other: Laboratory Biomarker Analysis — Correlative Studies
Procedure: Surgical Procedure — Undergo surgical tumor resection
  Other Names: Operation; Surgery; Surgical; Surgical Interventions; Surgical Procedures
Biological: Tremelimumab — Given IV
  Other Names: Anti-CTLA4 Human Monoclonal Antibody CP-675,206; CP-675; CP-675,206; CP-675206; Ticilimumab
  Arms: Treatment (tremelimumab and durvalumab); Treatment (tremelimumab)

SUMMARY:
The main purpose of this trial is to investigate the effects of a new class of drugs that help the patient's immune system attack their tumor (glioblastoma multiforme - GBM). These drugs have already shown benefit in some other cancer types and are now being explored in GBM. Both tremelimumab and durvalumab (MEDI4736) are "investigational" drugs, which means that the drugs are not approved by the Food and Drug Administration (FDA). Both drugs are antibodies (proteins used by the immune system to fight infections and cancers). Durvalumab attaches to a protein in tumors called PD-L1. It may prevent cancer growth by helping certain blood cells of the immune system get rid of the tumor. Tremelimumab stimulates (wakes up) the immune system to attack the tumor by inhibiting a protein molecule called CTLA-4 on immune cells. Combining the actions of these drugs may result in better treatment options for patients with glioblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the T-cell changes that occur in glioblastoma (GBM) treated with tremelimumab and durvalumab (MEDI4736) as single agents and in combination.

SECONDARY OBJECTIVES:

I. To evaluate the safety of either tremelimumab or MEDI4736 alone and in combination in patients with GBM.

II. To determine the time to progression for patients treated with either tremelimumab or MEDI4736 alone and in combination of both, post-surgery.

III. To determine the overall survival for patients treated with tremelimumab or MEDI4736 alone and in combination of both post-surgery.

IV. To assess magnetic resonance imaging (MRI) changes in patients treated with either tremelimumab or MEDI4736 alone and in combination of both post-surgery.

TERTIARY OBJECTIVES:

I. To correlate T-cell changes and programmed death ligand 1 (PDL1) expression with patient outcomes.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM 1: Patients receive tremelimumab intravenously (IV) over 1 hour on day 1. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

ARM 2: Patients receive durvalumab IV over 1 hour on days 1 and 15. Courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity.

ARM 3: Patients receive tremelimumab IV over 1 hour on day 1 then, after a gap of 1 hour for the first cycle, durvalumab IV over 1 hour on days 1 and 15. Courses repeat every 4 weeks with tremelimumab for up to 7 courses and every 2 weeks with durvalumab for up to 14 courses. Patients then receive both tremelimumab and durvalumab IV over 1 hour every 12 weeks in the absence of disease progression or unacceptable toxicity.

All patients undergo surgical tumor resection on day 14.

After completion of study treatment, patients are followed up every 8-16 weeks for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a grade III or IV glioma that has progressed after standard radiotherapy (RT) and temozolomide (TMZ) (Note: Pathology will need to be reviewed locally but registration can occur based on pathology report)
* Patients must have had radiographic evidence of tumor progression by brain MRI or computed tomography (CT) scan with contrast
* Patients must be > 12 weeks from completion of radiation therapy unless there is tissue confirmation of tumor recurrence or there is progression outside the radiation treatment field
* Prior therapy with gamma knife or other focal high-dose radiotherapy is allowed, but the patient must have subsequent histologic documentation of recurrence, unless the recurrence occurs remote from the treated site
* Patients must be surgical candidates
* Patients must have had no more than 3 prior lines of chemotherapy; this includes the initial treatment and two relapses; concurrent and adjuvant TMZ-based chemotherapy, including the combination of TMZ with another agent, is considered one line of chemotherapy; for clarification, please contact the principle investigator (PI), Dr. Jeffrey Raizer, at (312) 695-0990
* Patients must be >=

  * 4 weeks from TMZ
  * 6 weeks from a nitrosoureas
  * 3 weeks from a biologic or targeted agent (i.e. small molecule)
  * 4 weeks for a vascular endothelial growth factor (VEGF) inhibitor (i.e. bevacizumab)
* Patients must exhibit a Karnofsky performance status (KPS) >= 70
* Life expectancy of >= 12 weeks (per treating investigator's discretion)
* Patients must be on a stable or decreasing dose of corticosteroids within 5 days prior to CT scan or MRI (which is done to determine eligibility); the goal should be dexamethasone 4 mg or less at the time of starting treatment; if patient requires > 4mg of steroid, please check with the principle investigator (PI); requirement for greater than 10mg of steroid will make the patient ineligible
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcl
* Hemoglobin (Hb) > 10.0 g/dL (can be transfused to this level)
* International Normalized Ratio (INR), prothrombin time (PT), or activated partial thromboplastin time (aPTT) as follows:

  * In the absence of therapeutic intent to anticoagulate the patient: INR < 1.5 or PT < 1.5 x upper normal limit (ULN) or aPTT < 1.5 x ULN
  * In the presence of therapeutic intent to anticoagulate the patient: INR or PT and aPTT within therapeutic limits (according to the medical standard in the institution) and the patient has been on a stable dose of anticoagulants for at least 2 weeks before registration
* Total bilirubin =< 1.5 x ULN (except in patients with Gilbert's disease)
* Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT)/ alanine aminotransferase (ALT) serum glutamic pyruvic transaminase (SPGT) =< 2.5 X institutional upper limit of normal (ULN)
* Serum creatinine < 1.5 x ULN
* Serum creatinine clearance (CL) > 40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance
* Females of child-bearing potential (FOCBP) and males must agree to use adequate contraception (e.g. hormonal or barrier method of birth control prior to registration, for the duration of study participation, and for 180 days after the last dose of MEDI4736 + tremelimumab combination therapy or 90 days after the last dose of MEDI4736 or tremelimumab monotherapy; should a female patient become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately

NOTE: A FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets both of the following criteria:

* Has not undergone a hysterectomy or bilateral oophorectomy
* Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)

  * FOCBP must have a negative pregnancy test (serum or urine) within 7 days prior to registration on study
  * Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study
  * Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up
  * Malignancy treated with curative intent and with no known active disease >=3 years before the first dose of study drug and of low potential risk for recurrence; NOTE: the exceptions to this requirement include adequately treated non-melanoma skin cancer or lentigo maligna or carcinoma in situ without evidence of disease
  * Patients can only be on non-enzyme inducing anti-convulsants; if they are on an enzyme inducing anti-convulsant, they may be converted to a non-enzyme inducing anti-convulsants but they will need a 2 week wash out period from time of drug discontinuation until day 1 of study treatment
  * Patients must have given written, signed and dated informed consent prior to registration on the study; NOTE: no study-specific screening procedures may be performed until consent has been given

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site); previous enrolment or randomization in the present study
* Has received prior therapy with an anti-programmed cell death protein 1 (PD-1), anti-programmed cell death ligand 2 (PD-L2), anti-cluster of differentiation (CD)137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
* Has known active hepatitis B (e.g., hepatitis B virus antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis c virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Known active human immunodeficiency virus (HIV1/2 antibodies)
* Patient has history of primary immunodeficiency OR has received any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment, excluding intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses; attempts should be made to have patient on lowest possible dose of steroids (acceptable range 4-10mg, please contact PI if dose is >4 mg) and weaned to off as is feasible
* Patients receiving any other investigational chemotherapeutic agents within 30 days prior to the first dose of trial treatment
* Mean QT interval corrected for heart rate (QTc) >= 470 ms calculated from an electrocardiograms (ECGs) using Bazett's Correction; if first ECG is abnormal, then the mean will be calculated from 3 consecutive ECGs (taken 2-5 minutes apart); please contact the PI for further clarification
* Active or prior documented history of immunologic disorder including autoimmune disease within the past 2 years NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
* History of allogeneic organ transplant
* Uncontrolled intercurrent illness including, but not limited to,

  * Ongoing or active infection,
  * Symptomatic congestive heart failure,
  * Uncontrolled hypertension (defined as > 150/90)
  * Unstable angina pectoris,
  * Cardiac arrhythmia,
  * Active peptic ulcer disease or gastritis,
  * Active bleeding diatheses
  * Psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
* Known history of previous clinical diagnosis of tuberculosis
* History of leptomeningeal carcinomatosis
* Receipt of live attenuated vaccination within 30 days prior to study entry (or due to receive one within 30 days of receiving either MEDI4736 or tremelimumab)
* Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
* Subjects with uncontrolled seizures
* Patients who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to MEDI3475 are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-05-09 (Actual); Study Completion 2020-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Raizer, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to accrual on September 13th, 2016 with an accrual goal of 36 patients. The first patient was enrolled onto the study and started treatment on November 1st, 2016. The accrual goal was met on April 5th, 2018. The study intended to increase the accrual goal, but the funding sponsor did not approve additional funding. The study closed permanently to further enrollment of participants on January 22nd, 2019.
Groups:
- Arm 1: Tremelimumab Only: * Pre-Surgery (14 days +/-3 days prior to surgery): One dose of tremelimumab IV, 75 mg.
  * Post-surgical MRI of brain will be done 72 hours after surgery.
  * Post-Surgery (14 days after surgery): Tremelimumab IV, 5 mg, every 4 weeks for up to 24 months until disease progression or unacceptable toxicity.
  * Contrast-enhanced MRI or CT scan will be done approximately every 2 cycles or 8 weeks.
- Arm 2: MEDI4736 Only: * Pre-Surgery (14 days +/-3 days prior to surgery): One dose of MEDI4736, 750 mg IV
  * Post-surgical MRI of brain will be done within 72 hours after surgery.
  * Post-Surgery (14 days after surgery): MEDI4736, 750 mg IV every 2 weeks for up to 24 months until disease progression or unacceptable toxicity.
  * Contrast-enhanced MRI or CT scan will be done approximately every 2 cycles or 8 weeks
- Arm 3: Tremelimumab + MEDI4736: * Pre-Surgery (14 days +/-3 days prior to surgery): One dose of tremelimumab IV, 75 mg, one dose of MEDI4736, 750 mg IV
  * Post-surgical MRI of brain will be done within 72 hours after surgery.
  * Post-Surgery (14 days after surgery): Tremelimumab IV, 75 mg, every 4 weeks (for up to 7 doses), MEDI4736 IV, 750 mg, every 2 weeks (for up to 14 doses).
  * Starting C7D1 (week 25): Tremelimumab IV, 75 mg, every 12 weeks and MEDI4736 IV, 750mg, every 2 weeks, for up to 24 months until disease progression or unacceptable toxicity.
  * On days when tremelimubab and MEDI4736 are given on the same day, tremilimumab is administered first, then MED14736 infused after a gap of 1 hour for the first cycle. If tolerated, then can be given one after the other for subsequent infusions.
  * Contrast-enhanced MRI or CT scan will be done approximately every 2 cycles or 8 weeks
Period: Pre-Surgical Treatment
Arm/Group | Arm 1: Tremelimumab Only | Arm 2: MEDI4736 Only | Arm 3: Tremelimumab + MEDI4736
Started | 12 | 12 | 12
Registered for Study | 12 | 12 | 12
Received First Dose (Pre-surgical Dose) of Study Drug | 12 | 11 | 11
Completed | 12 | 11 | 11
Not Completed | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Progressive Disease | 0 | 1 | 0
Period: Post-Surgery Treatment (Adjuvant)
Arm/Group | Arm 1: Tremelimumab Only | Arm 2: MEDI4736 Only | Arm 3: Tremelimumab + MEDI4736
Started | 12 | 11 | 11
Started Cycle 1 | 11 | 8 | 11
Started Cycle 2 | 7 | 8 | 11
Started Cycle 3 | 3 | 7 | 4
Started Cycle 4 | 2 | 5 | 2
Started Cycle 5 | 2 | 3 | 2
Started Cycle 6 | 0 | 3 | 2
Started Cycle 7 | 0 | 3 | 1
Started Cycle 8 | 0 | 3 | 1
Started Cycle 9 | 0 | 3 | 1
Started Cycle 10 | 0 | 2 | 1
Started Cycle 11 | 0 | 2 | 1
Started Cycle 12 | 0 | 1 | 1
Started Cycle 13 | 0 | 1 | 1
Started Cycle 14 | 0 | 1 | 1
Started Cycle 15 | 0 | 0 | 1
Started Cycle 16 | 0 | 0 | 1
Started Cycle 17 | 0 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 12 | 11 | 11
Not completed — Withdrawal by Subject | 1 | 4 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Progressive Disease | 10 | 6 | 10
Not completed — Adverse Event | 0 | 1 | 1
Period: Follow-up Period (up to 2 Years)
Arm/Group | Arm 1: Tremelimumab Only | Arm 2: MEDI4736 Only | Arm 3: Tremelimumab + MEDI4736
Started (All patients who receive at least 1 dose of study drug go into follow-up.) | 12 | 11 | 11
Completed | 0 | 1 | 1
Not Completed | 12 | 10 | 10
Not completed — Death | 12 | 10 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Tremelimumab Only | Arm 2: MEDI4736 Only | Arm 3: Tremelimumab + MEDI4736 | Total
Number analyzed (Participants) | 12 | 12 | 12 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 8 | 29
  >=65 years | 1 | 2 | 4 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 5 | 12
  Male | 8 | 9 | 7 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 1 | 5
  Not Hispanic or Latino | 9 | 11 | 11 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 10 | 11 | 12 | 33
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 12 | 36

OUTCOME MEASURES:

1. Primary Outcome: T-cell (Immunologic) Changes in Blood
Description: To determine the T-cell changes that occur in glioblastoma treated with tremelimumab and MEDI4736 as single agents and in combination. The changes from baseline will be assessed in blood samples and tissue samples before pre-surgery treatment with MEDI4736 and/or tremelimumab, day of surgery, and during adjuvant treatment, for all patients in the 3 arms.
Time Frame: From baseline up to end of treatment, where all patients received at least 1 dose pre-surgery, and range of cycles attempted post-surgery was 0-16 (1 Cycle = 4 weeks)
Population: Blood samples were collected from patients and shipped to an outside organization. The PI has contacted the outside organization to request T-cell data to be collected from blood samples and followed up multiple times. Outside organization has been unresponsive. There is no data collected from blood samples and will not be any data generated in the future from bloods samples for this endpoint. We have no data to report for this endpoint
Arm/Group | Arm 1: Tremelimumab Only | Arm 2: MEDI4736 Only | Arm 3: Tremelimumab + MEDI4736
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: MRI Changes
Description: To assess MRI changes in lesion size in patients treated with either Tremelimumab or MEDI4736 alone and in combination of both post surgery. Only patients who have been administered at least one dose of investigational drug, undergone surgery, and have undergone at least one post-surgery disease assessment will be evaluable for this endpoint. Changes will be summarized using means. MRI changes below show the changes from baseline to after surgery.
Time Frame: Baseline and 3 days after surgery
Measure: Mean (Standard Deviation); unit: milimeters squared
Arm/Group | Arm 1: Tremelimumab Only | Arm 2: MEDI4736 Only | Arm 3: Tremelimumab + MEDI4736
Number analyzed (Participants) | 11 | 9 | 11
milimeters squared | 1410 (4290) | 1720 (2730) | 3020 (7320)

3. Secondary Outcome: Number of Patients Adverse Events Regardless of Attribution to the Study Drug Graded 3, 4, and 5
Description: Toxicity, both frequency and severity, will continue to be measured by monitoring the occurrence of adverse events. Adverse events will be defined as those included in CTCAE v 4.03. AEs graded 3, 4, 5 (regardless of attribution to the study drug) are included here. Grade 1 (mild): the event causes discomfort without disruption of normal daily activities. Grade 2 (moderate): the event causes discomfort that affects normal daily activities. Grade 3 (severe): the event makes the patient unable to perform normal daily activities or significantly affects his/her clinical status. Grade 4 (Life-threatening): the patient was at risk of death at the time of the event. Grade 5 (fatal): the event caused death.
Time Frame: From baseline, pre-surgery treatment period (2 weeks prior to surgery), and post-surgery treatement, where the range of cycles attempted post-surgery was 0-16 (1 Cycle = 4 weeks), to 90 days post treatment discontinuation
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Tremelimumab Only | Arm 2: MEDI4736 Only | Arm 3: Tremelimumab + MEDI4736
Number analyzed (Participants) | 12 | 11 | 11
Participants
  Grade 5 Disease Progression | 5 | 4 | 2
  Grade 3 Left-sided Weakness | 1 | 0 | 1
  Grade 3 UTI | 2 | 0 | 1
  Grade 3 Pulmonary Embolism | 1 | 0 | 0
  Grade 3 Fall | 1 | 0 | 0
  Grade 5 Intracranial hemorrhage | 1 | 0 | 0
  Grade 4 Encephalopathy | 1 | 1 | 0
  Grade 4 Seizures | 1 | 0 | 0
  Grade 3 Seizures | 1 | 4 | 2
  Grade 3 Clinical decline | 2 | 0 | 0
  Grade 3 Acute Encephalopathy | 1 | 0 | 0
  Grade 3 Viral meningitis | 0 | 1 | 0
  Grade 3 Back Pain | 0 | 1 | 0
  Grade 3 Weakness | 0 | 1 | 0
  Grade 3 Encephalopathy | 0 | 1 | 1
  Grade 3 Intraparenchymal hemorrhage | 0 | 1 | 0
  Grade 3 Hydrocephalus | 0 | 1 | 0
  Grade 3 Gait imbalance | 0 | 1 | 0
  Grade 3 Colitis | 0 | 0 | 1
  Grade 4 Sepsis | 0 | 0 | 1
  Grade 3 Wound Infection | 0 | 0 | 1
  Grade 3 Stroke | 0 | 0 | 1
  Grade 3 Wound dehiscence | 0 | 0 | 1

4. Secondary Outcome: Overall Survival
Description: To determine post-surgery the overall survival for patients treated with Tremelimumab or MEDI4736 alone and in combination. This will be defined as the number of months surviving from the time of first dose of study treatment until death by any cause. Only patients who have been administered at least one dose of investigational drug and undergone surgery will be evaluable for this endpoint.
Time Frame: From the start of treatment (pre-surgery treatment period = 2 weeks), to surgery, to post-surgery treatment, where range of cycles attempted was 0-16 (1 Cycle = 4 weeks), to 2 years post treatment discontinuation
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1: Tremelimumab Only | Arm 2: MEDI4736 Only | Arm 3: Tremelimumab + MEDI4736
Number analyzed (Participants) | 11 | 9 | 11
months | 7.246 [2.746 to 16.32] | 11.71 [8.332 to 32.71] | 7.703 [7.411 to 40.14]

5. Secondary Outcome: Time to Progression
Description: To the time to progression (per Modified RANO criteria and iRANO criteria) for patients treated with either Tremelimumab or MEDI4736 alone and in combination. This will be defined as the number of months from the time of first dose of study treatment until progression of disease (PD) or death from any cause. Only patients who have been administered at least one dose of investigational drug and undergone surgery will be evaluable for this endpoint. Definition of PD per RANO criteria: New contrast-enhancing lesion outside of radiation field on decreasing, stable, or increasing doses of corticosteroids; Increase by > 50% (modified from >25% according to published RANO criteria) enhancement from the first post-surgical scan, or a subsequent scan with smaller tumor size, and the scan 8 weeks or later on stable or increasing doses of corticosteroids; Clinical deterioration not attributable to concurrent medication or comorbid conditions.
Time Frame: From start of treatment (pre-surgery treatment period = 2 weeks), to surgery, to post-surgery treatment where range of cycles attempted was 0-16 (1 Cycle = 4 weeks), and up to 2 years of follow-up after treatment discontinuation
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1: Tremelimumab Only | Arm 2: MEDI4736 Only | Arm 3: Tremelimumab + MEDI4736
Number analyzed (Participants) | 11 | 9 | 11
months | 2.746 [2.68 to 8.727] | 4.356 [2.941 to 32.74] | 4.913 [2.905 to 120.4]

6. Other Pre Specified Outcome: T-cell Changes
Description: Immunologic changes of T-cells will be correlated to survival outcomes. T-cell changes will be measured from blood samples.
Time Frame: Up to 2 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: PDL1 Expression
Description: Immunologic changes of PDL1 levels will be correlated to survival outcomes. PDL1 levels will be measured from blood samples.
Time Frame: Up to 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected over a 3 year period. For other AEs ,each patient was followed from the time of treatment, during treatment at the beginning of each cycle through 90 days post last treatment. For Serious AEs, each patient was followed at time of consent and 90 days post last treatment. Patients received a single dose of study treatment pre-surgery. The range of adjuvant/post-surgery cycles attempted was 0-16 (1 cycle = 4 weeks).
Description: All cause mortality and other adverse events are assessed from first dose of study treatment. Only patients that received at least 1 dose of study drug are included in all cause mortality and other adverse events. SAEs are assessed from patient signing consent.
Arm/Group | Arm 1: Tremelimumab Only | Arm 2: MEDI4736 Only | Arm 3: Tremelimumab + MEDI4736
All-Cause Mortality (participants affected / at risk) | 12/12 | 10/11 | 10/11
Serious Adverse Events (participants affected / at risk) | 9/12 | 10/12 | 8/12
Other Adverse Events (participants affected / at risk) | 12/12 | 11/11 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Tremelimumab Only (N=12) | Arm 2: MEDI4736 Only (N=12) | Arm 3: Tremelimumab + MEDI4736 (N=12)
Seizures (Nervous system disorders) | 2 | 5 | 2 — 1 patient (in Arm 1) also experienced confusion. 1 patient (in Arm 2) also experienced headaches, nausea, and vomiting.
Disease Progression (General disorders) | 3 | 7 | 2
Left-sided weakness (Nervous system disorders) | 1 | 0 | 0
Urinary tract infection (Renal and urinary disorders) | 1 | 1 | 1 — One patient (in Arm 1) also experienced dyspnea. One patient (in Arm 3) also experienced left-sided weakness.
Pulmonary embolism (Vascular disorders) | 1 | 0 | 0 — One patient (in Arm 1) also experienced a fall.
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Intracranial hemorrhage (Nervous system disorders) | 1 | 0 | 0 — 1 patient (in Arm 1) also experienced a fall.
Encephalopathy (Nervous system disorders) | 1 | 3 | 1
Clinical decline (General disorders) | 0 | 2 | 1
Agitation (Psychiatric disorders) | 0 | 1 | 0
Mental status change (Nervous system disorders) | 0 | 1 | 0 — 1 patient (in Arm 2) also experienced a urinary tract infection.
Viral meningitis (Infections and infestations) | 0 | 1 | 0 — 1 patient (in Arm 2) also experienced a seizure.
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Weakness (Nervous system disorders) | 0 | 2 | 0
Intraparenchymal hemorrhage (Nervous system disorders) | 0 | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1 | 0
Gait imbalance (General disorders) | 0 | 1 | 0
Nausea/Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 — 1 patient (in Arm 3) also experienced clinical decline.
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 — 1 patient (in Arm 3) also experienced acute kidney injury.
Wound infection (Infections and infestations) | 0 | 0 | 1
Stroke (Nervous system disorders) | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Tremelimumab Only (N=12) | Arm 2: MEDI4736 Only (N=11) | Arm 3: Tremelimumab + MEDI4736 (N=11)
Anemia (Blood and lymphatic system disorders) | 7 | 9 | 9
Blood and lymphatic disorders NOS (Blood and lymphatic system disorders) | 0 | 0 | 2
Palpatations (Cardiac disorders) | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 4 | 3 | 2
Sinus tachycardia (Cardiac disorders) | 2 | 5 | 2
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 1 | 1
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 2
Cushingoid (Endocrine disorders) | 1 | 0 | 0
Thyroiditis (Endocrine disorders) | 0 | 0 | 1
Blurred vision (Eye disorders) | 0 | 1 | 0
Eyelid function disorder (Eye disorders) | 1 | 0 | 0
Esotropia (Eye disorders) | 0 | 1 | 0
Optic nerve disorder (Eye disorders) | 0 | 0 | 2
Ptosis (Eye disorders) | 0 | 1 | 0
Quadrantanopsia (Eye disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 1 | 3
Diarrhea (Gastrointestinal disorders) | 3 | 3 | 2
Dry throat (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Fecal incontinence (Gastrointestinal disorders) | 1 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 3 | 1 | 4
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Chills (General disorders) | 0 | 1 | 2
Edema limbs (General disorders) | 0 | 1 | 0
Facial pain (General disorders) | 1 | 0 | 1
Fatigue (General disorders) | 5 | 2 | 7
Fever (General disorders) | 1 | 4 | 1
Gait disturbance (General disorders) | 4 | 2 | 1
Irritability (General disorders) | 1 | 0 | 0
Localized edema (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 3
Facial droop (General disorders) | 0 | 1 | 0
Leg Swelling (General disorders) | 0 | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 1 | 0
Transaminitis (General disorders) | 0 | 1 | 0
Infusion related reaction (General disorders) | 0 | 1 | 0
Oral thrush (Infections and infestations) | 0 | 1 | 0
Staph infection (Infections and infestations) | 0 | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0
Chest congestion (Infections and infestations) | 1 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 2 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 1
Activated partial thromboplastin time prolonged (Investigations) | 2 | 0 | 1
Alanine aminotransferase increased (Investigations) | 3 | 3 | 3
Alkaline phosphatase increased (Investigations) | 6 | 3 | 5
Aspartate aminotransferase increased (Investigations) | 2 | 3 | 3
Blood bilirubin increased (Investigations) | 2 | 1 | 2
Creatinine increased (Investigations) | 1 | 2 | 1
Fibrinoigen decreased (Investigations) | 0 | 0 | 1
INR increased (Investigations) | 0 | 1 | 2
Lymphocyte count decreased (Investigations) | 8 | 8 | 9
Neutrophil count decreased (Investigations) | 1 | 2 | 1
Platelet count decreased (Investigations) | 3 | 6 | 7
Weight gain (Investigations) | 3 | 1 | 0
Weight loss (Investigations) | 0 | 4 | 1
White blood cell decreased (Investigations) | 2 | 2 | 4
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 2
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 11 | 11 | 10
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Hypernatremia (Metabolism and nutrition disorders) | 3 | 1 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 | 6 | 9
Hypocalcemia (Metabolism and nutrition disorders) | 4 | 2 | 4
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 4 | 7 | 7
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 5
Hyponatremia (Metabolism and nutrition disorders) | 3 | 4 | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 5 | 5 | 6
Mixed hyperlipidemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Steroid myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Shoulder pain (intermittent) (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
pseudomeningocele (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
epidural hematoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 0
Ataxia (Nervous system disorders) | 5 | 1 | 0
Cognitive disturbance (Nervous system disorders) | 2 | 1 | 3
Concentration impairment (Nervous system disorders) | 1 | 2 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1
Dysarthria (Nervous system disorders) | 1 | 2 | 0
Dysesthesia (Nervous system disorders) | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 1
Dysphasia (Nervous system disorders) | 2 | 1 | 1
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Facial muscle weakness (Nervous system disorders) | 3 | 0 | 1
Headache (Nervous system disorders) | 7 | 7 | 3
Hypersomnia (Nervous system disorders) | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0
Paraphasia (Nervous system disorders) | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 2 | 4 | 2
Sleep disturbance (Nervous system disorders) | 0 | 0 | 1
Expressive aphasia (Nervous system disorders) | 0 | 0 | 1
Paresthesia (Nervous system disorders) | 0 | 0 | 1
Coma (Nervous system disorders) | 0 | 1 | 0
Disorientation (Nervous system disorders) | 0 | 1 | 0
Intermittent slurred speech (Nervous system disorders) | 0 | 1 | 0
Hemineglect (Nervous system disorders) | 0 | 1 | 0
Left sided hemiparesis (Nervous system disorders) | 0 | 1 | 0
Proprioception difficulties (Nervous system disorders) | 0 | 1 | 0
Aphasia (Nervous system disorders) | 2 | 0 | 0
Intercranial edema (Nervous system disorders) | 1 | 0 | 0
Pronator drift (Nervous system disorders) | 2 | 1 | 0
Nystagmus (Nervous system disorders) | 0 | 1 | 0
Oculomotor nerve disorder (Nervous system disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 3 | 1 | 2
Spasticity (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 1
Confusion (Psychiatric disorders) | 3 | 5 | 2
Depression (Psychiatric disorders) | 0 | 1 | 1
Hallucinations (Psychiatric disorders) | 1 | 2 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 0
Abulia (Psychiatric disorders) | 1 | 0 | 0
Anhedonia (Psychiatric disorders) | 1 | 0 | 0
Tearful (Psychiatric disorders) | 1 | 0 | 0
Hematuria (Renal and urinary disorders) | 1 | 1 | 2
Proteinuria (Renal and urinary disorders) | 1 | 1 | 2
Nocturnal Urination (Renal and urinary disorders) | 0 | 1 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 3 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 2 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oral mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acute bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
Psoriatic flair (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 11 | 7 | 8
Hypotension (Vascular disorders) | 0 | 0 | 2
Thromboembolic event (Vascular disorders) | 0 | 3 | 0
Change in temperature (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/83/NCT02794883/Prot_SAP_000.pdf